CLINICAL TRIAL: NCT00717522
Title: A Phase 2, Multicenter, Open-label, Single Arm, Two-stage Study to Evaluate the Efficacy and Safety of CC-4047 (Pomalidomide) in Patients With Advanced Soft Tissue Sarcomas Who Have Relapsed or Are Refractory to Systemic Anticancer Therapy
Brief Title: Efficacy and Safety Study of CC-4047 (Pomalidomide) to Treat Advanced Soft Tissue Sarcoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study enrollment was terminated due to a corporate strategic decision unrelated to patient safety.
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-4047-STSAR-001
Record Dates: First submitted 2008-07-16; First posted 2008-07-17 (Estimated); Results first posted 2013-04-16 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Soft Tissue Sarcoma
Keywords: Soft Tissue Sarcoma; CC-4047; Pomalidomide
MeSH Terms: conditions — Sarcoma | interventions — pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pomalidomide (Experimental): 7 mg pomalidomide taken orally once daily (QD) on days 1 through 21 of each 28-day cycle
  Interventions: Drug: Pomalidomide

INTERVENTIONS:
Drug: Pomalidomide
  Other Names: CC-4047; Pomalyst

SUMMARY:
The purpose of the study is to determine the safety and efficacy of single agent CC-4047 (pomalidomide) in patients with advanced soft tissue sarcomas who have relapsed or are refractory to prior anticancer therapy.

ELIGIBILITY:
Inclusion Criteria:

* Must be > 18 years of age
* Must have histologically confirmed soft tissue sarcoma
* Must have locally recurrent unresectable, or metastatic soft tissue sarcoma, and have failed or relapsed after a minimum of one and a maximum of 3 prior systemic anticancer therapy regimens
* Must have measurable or evaluable disease determined as per Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Must have documented disease progression (PD) determined as per RECIST criteria within 3 months prior to study enrollment
* Must have Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1

Exclusion Criteria:

* Pregnant or lactating females
* Prior therapy with thalidomide or lenalidomide
* Prior use of experimental/investigational drug therapy < 3 months prior to treatment initiation
* Prior chemotherapy, biologic or immunotherapy < 3 weeks prior to treatment initiation
* Prior radiotherapy < 3 weeks prior to treatment initiation
* Prior major surgery < 3 weeks prior to treatment initiation
* Absolute neutrophil count (ANC) < 1.5 x 109 cells/L
* Platelet count < 100 x 109cells/L
* Aspartate aminotransferase/serum glutamic oxaloacetic transaminase (AST/SGOT) and alanine aminotransferase/serum glutamic pyruvate transaminase (ALT/SGPT) > 3.0 x upper limit of normal (ULN) or > 5.0 x ULN in the presence of demonstrable liver metastases
* Known active central nervous system (CNS) metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-08-01 (Actual); Primary Completion 2009-01-01 (Actual); Study Completion 2009-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abderrahim Fandi, MD, Study Director — Celgene
Locations (3):
- United States (3):
  - Sarcoma Oncology Center, Santa Monica, California
  - Kootenai Cancer Center, Coeur d'Alene, Idaho
  - Nebraska Methodist Hospital, Omaha, Nebraska

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pomalidomide
Started | 7
Completed | 0
Not Completed | 7
Not completed — Disease Progression | 5
Not completed — Adverse Event | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pomalidomide
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (13.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Race/Ethnicity, Customized [Number; unit: participants]
  White | 7
  Non-white | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Deaths, or Discontinuations Due to AEs
Description: An adverse event (AE) is defined as any noxious, unintended, or untoward medical occurrence occurring at any dose that may appear or worsen in a study subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the study subject's health, including laboratory test values, regardless of etiology. A serious adverse event (SAE) is defined as any AE which: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; constitutes an important medical event. National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE), Version 3.0, grades: 1 = mild, 2 = moderate, 3 = severe, 4 = life threatening, 5 = death. For more details, please see the Adverse Events section of this record.
Time Frame: AEs/SAEs were recorded from informed consent to 30 days post treatment discontinuation visit. Median treatment duration was 49 days (range: 3 to 102 days).
Population: All participants
Measure: Number; unit: participants
Arm/Group | Pomalidomide
Number analyzed (Participants) | 7
participants
  ≥1 AE | 7
  ≥1 AE suspected to be related to study drug | 6
  ≥1 Grade 3 AE | 4
  ≥1 Grade 4 AE | 1
  ≥1 SAE | 3
  ≥1 SAE suspected to be related to study drug | 1
  Death | 4
  Death within 30 days of last dose of study drug | 1
  Discontinuation due to AE | 2
  Dose reduction and interruption due to AE | 1

2. Secondary Outcome: Tumor Response as Assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee Guidelines
Description: Changes in only the longest diameter (LD) of tumor lesions are used in RECIST criteria. Evaluation of target lesions: Complete Response (CR)=Disappearance of all target lesions; Partial Response (PR)=≥30% decrease in sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD; Progressed Disease (PD)=≥20% increase in sum of LD of target lesions taking as reference the smallest sum LD recorded since treatment started or the appearance of ≥1 new lesions; Stable Disease (SD)=Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as reference the smallest sum LD since treatment started. For non-target lesions: CR= Disappearance of all non-target lesions and normalization of tumor marker level; Incomplete Response/SD=Persistence of ≥1 non-target lesions and/or maintenance of tumor marker level above normal limits; PD=Appearance of ≥1 new lesions; unequivocal progression of existing non-target lesions.
Time Frame: Assessed every 8 weeks for the first 8 months and then every 12 weeks thereafter, and at treatment discontinuation. Median treatment duration was 49 days (range: 3 to 102 days).
Population: This analysis was not done. Study enrollment was suspended due to a corporate strategic decision unrelated to patient safety, and the protocol was amended to evaluate safety only (efficacy data was stored but not cleaned or analyzed unless related to safety).
Arm/Group | Pomalidomide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) are defined as any AE occurring or worsening on or after the first treatment of the study medication and within 30 days after the last dose. Median treatment duration was 49 days (range: 3 to 102 days).
Arm/Group | Pomalidomide
Serious Adverse Events (participants affected / at risk) | 3/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pomalidomide (N=7)
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Sarcoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Tachycardia (Cardiac disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1
Syncope (Nervous system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pomalidomide (N=7)
Nausea (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Palatal disorder (Gastrointestinal disorders) | 1
Tongue disorder (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Asthenia (General disorders) | 1
Chills (General disorders) | 1
Malaise (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Alanine aminotransferase increased (Investigations) | 1
Ammonia increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Electrocardiogram q waves (Investigations) | 1
International normalised ratio increased (Investigations) | 1
Weight decreased (Investigations) | 1
Dizziness (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Vocal cord paralysis (Nervous system disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Cachexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hypophagia (Metabolism and nutrition disorders) | 1
Iron deficiency (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Anxiety (Psychiatric disorders) | 1
Libido decreased (Psychiatric disorders) | 1
Personality change (Psychiatric disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Deep vein thrombosis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Upon investigator submission of a publication or presentation to Celgene, Celgene shall complete its review within 60 days after receipt of the proposed publication or presentation. Upon Celgene's request, proposed publication or presentation will be delayed up to 60 additional days to enable Celgene to secure adequate intellectual property protection of property of Celgene that would be affected by such proposed publication or presentation.